CLINICAL TRIAL: NCT00325832
Title: Conventional Versus Automated Measurement of Blood Pressure in the Office (The CAMBO Study)
Acronym: CAMBO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 392-2005
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure; Systolic Pressure; Diastolic Pressure; Blood Pressure Monitoring, Ambulatory
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BpTRU
Device: Conventional mercury sphygmomanometry

SUMMARY:
To determine if the use of automated office blood pressure readings can improve management of systolic hypertension in routine clinical practice. Automated office SBP recordings in routine clinical practice using the BpTRU device will reflect more accurately the mean awake ambulatory systolic BP than will manual BP readings taken with conventional mercury sphygmomanometry. This should lead to improvements in the management of systolic hypertension with optimization of drug therapy in practices using the BpTRU device.

ELIGIBILITY:
Inclusion Criteria:

* Both treated and untreated patients with systolic hypertension under routine FP care
* For untreated patients, routine office SBP as measured by the patient's FP at the last routine office visit using a mercury device must have SBP ≥ 160 mmHg and DBP <= 95 mmHg
* For patients already receiving antihypertensive therapy, the last routine office BP as measured by the patient's FP using mercury sphygmomanometry must be SBP ≥ 140 mmHg and DBP <= 90 mmHg

Exclusion Criteria:

* Presence of target organ damage such as MI, stroke, and serum creatinine twice normal
* Diabetes mellitus treated with insulin or oral hypoglycemic therapy
* Secondary hypertension
* Participation in another research study involving measurement of BP
* Patient's insistence on using self BP measurement outside of the study
* Any conditions or circumstances which might preclude the successful completion of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
ambulatory blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Martin Myers, MD, Principal Investigator — Sunnybrook Medical Sciences Centre; Sheldon Tobe, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada